CLINICAL TRIAL: NCT02438553
Title: A Prospective, Randomized, Single Blind, Parallel-group, Placebo Controlled Clinical Study to Evaluate the Short-term Effectiveness of Combined Occipital and Supraorbital Transcutaneous Nerve Stimulation (OS-TNS) in Reducing Migraine Related Pain
Brief Title: Short-term Effectiveness of Transcutaneous Nerve Stimulation in Reducing Migraine Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRLF-0086-14-MMC-CTIL
Record Dates: First submitted 2015-05-03; First posted 2015-05-08 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSTNS Neurostimulator (Experimental): Combined Occipital & Supraorbital Transcutaneous Neurostimulator.
  Interventions: Device: OSTNS Neurostimulator
- Placebo OSTNS Neurostimulator (Placebo Comparator): Placebo Combined Occipital & Supraorbital Transcutaneous Neurostimulator.
  Interventions: Device: Placebo OSTNS Neurostimulator

INTERVENTIONS:
Device: OSTNS Neurostimulator — Non-invasive transcutaneous neurostimulation.
  Other Names: Transcutaneous Neurostimulator.
  Arms: OSTNS Neurostimulator
Device: Placebo OSTNS Neurostimulator — Placebo non-invasive transcutaneous neurostimulation
  Other Names: Transcutaneous Neurostimulator
  Arms: Placebo OSTNS Neurostimulator

SUMMARY:
The purpose of this study is to evaluate the short-term effectiveness of combined occipital and supraorbital transcutaneous nerve stimulation in reducing migraine related pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of migraine headache without aura or with typical migraine with aura (ICHD-II code 1.2.1 or 1.1).
* Subjects with 1-6 migraine episodes per month in the last 2 months.
* The subject is capable of understanding the study and to sign an informed consent.

Exclusion Criteria:

* Subjects who have concomitant epilepsy.
* History of neurosurgical interventions.
* Subjects with metal implants or shrapnel in their head, except for dental implants.
* Subjects with implanted cardiac pacemaker, neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
* History of drug abuse or alcoholism.
* History of medications overuse headache.
* Participation in current clinical study or participated in a clinical study within 3 months prior to this study.
* Skin lesion or inflammation at the region of the stimulating electrodes.
* Personality or somatoform disorder.
* Pregnancy or Lactation.
* Women of reproductive age not using efficient contraceptive method.
* History of cerebrovascular event.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain visual analogue scale (VAS) | 20-60 minutes of treatment.
  The primary endpoint will be defined based on relative change (%) in pain VAS score from baseline to end of treatment without using pain relief medication.

SECONDARY OUTCOMES:
"Responder" rate at 20-60 minutes of treatment. | 20-60 minutes of treatment.
  - Evaluated using pain VAS; a responder will be defined by a decrease of 50% or more in the pain VAS from baseline to end of treatment without using pain relief medication.
"Responder" rate at 15 minutes of treatment | Baseline, 15 minutes of treatment
  Responder" rate at 15 minutes of treatment - Evaluated using pain VAS; a responder will be defined by a decrease of 50% or more in the pain VAS from baseline to end of treatment without using pain relief medication.
Sustained "Responder" rate at 24 hours post treatment | Baseline, 24 hours post treatment
  Sustained "responders" rate at 24 hours: The percentage of study participants who will be defined as a "responder" at 2 hour and will not use pain relief medication or suffer from relapse (recurrence) within the subsequent 24 hours.
"Headache relief" rate- at 2 hours | Baseline, 2 hours
  "Headache relief" rate- the percentage of subjects with a decrease in headache from severe or moderate to none or mild within 2 hours, before any pain relief medication.
Sustained "headache relief" at 24 hours | Baseline, 24 hours
  The percentage of study participants who will be defined as having a "headache relief" at 2 hour and will not use pain relief medication or suffer from relapse (recurrence) within the subsequent 24 hours.
Pain free at 2 hours | Baseline, 2 hours
  Percentage of subjects that are pain free at 2 hours
Sustained pain freedom at 24 hours | Baseline, 24 hours
  The percentage of study participants who will be defined as "pain free" at 2 hour and will not use pain relief medication or suffer from relapse (recurrence) within the subsequent 24 hours.
Functional disability change 2 hours from end of treatment | Baseline, 2 Hours post treatment
  Functional disability change 2 hours from end of treatment without using pain relief medication.
Time until use of pain relief medication. | Baseline- 24 hours.
  Time until use of pain relief medication.
Presence of nausea, vomiting, photophobia, phonophobia. | Baseline- 24 hours.
  Presence of nausea, vomiting, photophobia, phonophobia.
Percentage of subjects who completed the treatment. | Baseline-20 minutes of treatment
  Percentage of subjects who completed at least 20 minutes the treatment.
Global impression of effect | Baseline- 24 hours.
  Global impression of effect- A simple Likert-type verbal scale: very poor, poor, no opinion, good, very good.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hering, Dr., Principal Investigator — Director of headache clinic, Department of Neurology, Meir General Hospital, Kfar Saba, Israel.
Locations (1):
- Meir General Hospital, Kfar Saba, Israel

REFERENCES:
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Ahmed HE, White PF, Craig WF, Hamza MA, Ghoname ES, Gajraj NM. Use of percutaneous electrical nerve stimulation (PENS) in the short-term management of headache. Headache. 2000 Apr;40(4):311-5. doi: 10.1046/j.1526-4610.2000.00046.x. PMID 10759936
- [Background] Loder E. Triptan therapy in migraine. N Engl J Med. 2010 Jul 1;363(1):63-70. doi: 10.1056/NEJMct0910887. No abstract available. PMID 20592298
- [Background] Hann S, Sharan A. Dual occipital and supraorbital nerve stimulation for chronic migraine: a single-center experience, review of literature, and surgical considerations. Neurosurg Focus. 2013 Sep;35(3):E9. doi: 10.3171/2013.6.FOCUS13233. PMID 23991822
- [Background] Saper JR, Dodick DW, Silberstein SD, McCarville S, Sun M, Goadsby PJ; ONSTIM Investigators. Occipital nerve stimulation for the treatment of intractable chronic migraine headache: ONSTIM feasibility study. Cephalalgia. 2011 Feb;31(3):271-85. doi: 10.1177/0333102410381142. Epub 2010 Sep 22. PMID 20861241
- [Background] Schoenen J, Vandersmissen B, Jeangette S, Herroelen L, Vandenheede M, Gerard P, Magis D. Migraine prevention with a supraorbital transcutaneous stimulator: a randomized controlled trial. Neurology. 2013 Feb 19;80(8):697-704. doi: 10.1212/WNL.0b013e3182825055. Epub 2013 Feb 6. PMID 23390177
- [Background] Schwedt TJ. Occipital nerve stimulation for chronic migraine--interpreting the ONSTIM feasibility trial. Cephalalgia. 2011 Feb;31(3):262-3. doi: 10.1177/0333102410383591. Epub 2010 Sep 16. No abstract available. PMID 20847083
- [Background] Silberstein SD, Dodick DW, Saper J, Huh B, Slavin KV, Sharan A, Reed K, Narouze S, Mogilner A, Goldstein J, Trentman T, Vaisman J, Ordia J, Weber P, Deer T, Levy R, Diaz RL, Washburn SN, Mekhail N. Safety and efficacy of peripheral nerve stimulation of the occipital nerves for the management of chronic migraine: results from a randomized, multicenter, double-blinded, controlled study. Cephalalgia. 2012 Dec;32(16):1165-79. doi: 10.1177/0333102412462642. Epub 2012 Oct 3. PMID 23034698
- [Result] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463